CLINICAL TRIAL: NCT02888834
Title: Serious Adverse Drug Reaction and Their Preventability in the Elderly Over 65 Years
Brief Title: Serious Adverse Drug Reaction and Their Preventability
Acronym: SADR
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2015Ao008
Record Dates: First submitted 2016-08-19; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Adverse Drug Reaction
Keywords: elderly; adverse drug reactions; hospitalized subjects; community-dwelling
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Adverse Drug Reaction Reporting Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Adverse drug reaction: Patients aged over 65 years who presented a serious adverse drug reaction notified to the Regional Pharmacovigilance Center of Champagne-Ardenne between January and May 2013 were included in the study.
  Interventions: Other: Adverse drug reaction

INTERVENTIONS:
Other: Adverse drug reaction

SUMMARY:
Introduction: Elderly aged over 65 years accounted for around 17.5% of the French general population. Adverse drug reactions (ADR) are common in this population. In elderly subject, prevalence of ADRs ranged from 4.3% to 63.0%.

Aim: To describe the serious ADR in elderly subjects aged over 65 years and assess their preventability.

Methods: A retrospective study was conducted at the Regional Pharmacovigilance Center of Champagne-Ardenne (northeast of France) between January and May 2013. Patients aged over 65 years who presented a serious ADR notified to the Regional Pharmacovigilance Center were included in the study.

DETAILED DESCRIPTION:
Introduction: Elderly aged over 65 years accounted for around 17.5% of the French general population. Adverse drug reactions (ADR) are common in this population. In elderly subject, prevalence of ADRs ranged from 4.3% to 63.0%. Age itself is not a risk factor for ADRs but is a factor of severity of ADR. According to the World Health Organization (WHO), more than half of all ADRs are considered to be preventable in elderly subjects. They are most often the result of a mistake during the prescription phase, or the monitoring phase, or may be due to poor compliance or inappropriate self-medication. Drug prescription is based on guidelines derived from clinical trial that have not included elderly subject with multiple comorbidities. Data regarding drug safety from clinical trials alone are insufficient, hence the need to continue the monitoring of ADR after drug marketing.

Aim: To describe the serious ADR in elderly subjects aged over 65 years and assess their preventability.

Methods: A retrospective study was conducted at the Regional Pharmacovigilance Center of Champagne-Ardenne (northeast of France) between January and May 2013. Patients aged over 65 years who presented a serious ADR notified to the Regional Pharmacovigilance Center were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 65 years
* Patients who presented a serious adverse drug reaction notified to the Regional Pharmacovigilance Center of Champagne-Ardenne

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who presented an adverse drug reaction notified to the Regional Pharmacovigilance Center of Champagne-Ardenne.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The different type of serious ADR were coded according to Medical Dictionary for Regulatory Activities (MedDRA version 16.0) according to lowest-level terms (LLTs), and then grouped by system organ class (SOC). | 9 months

SECONDARY OUTCOMES:
Drugs involved in the occurrence of serious ADR | 9 months
Evolution were classified as "recovered", "not yet recovered", "recovered with sequelae" , "death" , "unknown" | 9 months
Preventability was assessed by using the preventability French scale. | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France

REFERENCES:
- [Background] Kanagaratnam L, Abou Taam M, Heng M, De Boissieu P, Roux MP, Trenque T. [Serious Adverse Drug Reaction and Their Preventability in the Elderly Over 65 Years]. Therapie. 2015 Sep-Oct;70(5):477-84. doi: 10.2515/therapie/2015029. Epub 2015 Jun 26. French. PMID 26223243